CLINICAL TRIAL: NCT01603953
Title: Malnutrition Assessed Through Bioelectrical Impedance Vector Analysis is Related to Poor Prognosis in Cirrhosis
Brief Title: Bioelectrical Impedance Vector Analysis in Cirrhotic Patients
Acronym: BIVA
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, ALDO TORRE DELGADILLO, M.D. M.Sc, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Other Study IDs: Gas-549-09-12-1
Record Dates: First submitted 2012-05-20; First posted 2012-05-23 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Cirrhosis; Hepatic Encephalopathy
MeSH Terms: conditions — Fibrosis; Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Protein-energy malnutrition and muscle wasting are a common finding among patients with liver cirrhosis. Its prevalence may range from 50-90% depending on the methods used for nutritional assessment. Even stable cirrhotic patients referred as Child A have muscle depletion and the majority of patients classified as Child C have significant depletion. Malnutrition has been shown to be related to several complications of cirrhosis

Despite the importance of nutritional status in patient's outcome, there is no gold standard for nutritional assessment. Traditional techniques used in healthy subjects to assess nutritional status cannot be used in cirrhotic patients due especially to ascites and peripheral edema, and altered rates of biochemical markers due to liver failure.

Bioelectrical impedance vector analysis has emerged as a useful method to assess body composition and nutritional status especially in patients at the extremes of body weight (fluid overload, excess of adipose tissue, etc.).

The aim of this study is to evaluate whether malnutrition assessed by bioelectrical impedance vector analysis is related to the development of hepatic encephalopathy

ELIGIBILITY:
Inclusion Criteria:

* Diagnose of cirrhosis.
* Ambulatory patients

Exclusion Criteria:

* Personal history of surgery in the last four weeks
* Thyroid disorders without replacement therapy
* Pregnancy
* Active alcoholism with alcohol ingest in the previous 6 months.
* Acute or chronic renal failure
* Hepatic or renal transplant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be recruited from the Gastroenterology Department of a tertiary care setting.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Hepatic encephalopathy | 6, 12, 24, 36 and 48 months
  Assessed by west Haven criteria

SECONDARY OUTCOMES:
Ascites | 6, 12, 24, 36 and 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Torre Delgadillo, M.D. M.Sc, Study Chair — INCMNSZ; Astrid Ruiz-Margáin, B.Sci, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico